CLINICAL TRIAL: NCT07349615
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase III Study to Evaluate the Efficacy and Safety of SHR-1918 in Patients With Hypertriglyceridemia
Brief Title: A Study of SHR-1918 In Participants With Hypertriglyceridemia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1918-305
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1918/ SHR-1918 placebo Group A , subcutaneous injection； (Experimental)
  Interventions: Drug: SHR-1918/ SHR-1918 placebo
- SHR-1918/ SHR-1918 placebo Group B, subcutaneous injection； (Experimental)
  Interventions: Drug: SHR-1918/ SHR-1918 placebo

INTERVENTIONS:
Drug: SHR-1918/ SHR-1918 placebo — SHR-1918/ SHR-1918 placebo Dose 1
  Arms: SHR-1918/ SHR-1918 placebo Group A , subcutaneous injection；
Drug: SHR-1918/ SHR-1918 placebo — SHR-1918/ SHR-1918 placebo Dose 2
  Arms: SHR-1918/ SHR-1918 placebo Group B, subcutaneous injection；

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of SHR-1918 in patients with hypertriglyceridemia. The efficacy and safety of SHR-1918 will be evaluated after 24-weeks and 48-weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ≥ 18 years old, who is able and willing to provide a written informed consent.
2. 1.7 ≤ TG ≤ 5.6 mmol/L.
3. LDL-C < 3.4 mmol/L.
4. Male and female subjects of childbearing potential and their partners must have no plans to donate sperm or become pregnant during the entire study period and after the last dose, and agree to use contraceptive methods as specified in the protocol.

Exclusion Criteria:

1. History of severe allergies/hypersensitivity reactions, or clinically significant allergies/hypersensitivity reactions as judged by the investigator, or history of allergies to drugs with similar chemical structures.
2. Received or are currently receiving treatment with monoclonal antibodies, siRNA-based drugs, or ASO-based drugs targeting the same target prior to screening.
3. Have a history of pancreatitis prior to screening or randomization.
4. Acute ischemic ASCVD events within 3 months prior to screening or randomization.
5. Heart failure with New York Heart Association (NYHA) Class III-IV prior to screening or randomization.
6. Malignant tumors within 5 years.
7. Received plasma exchange therapy within 2 months prior to screening, or plans to receive plasma exchange therapy during the study period, or has received LDL receptor gene therapy prior to screening.
8. Have a history of diseases that significantly affect blood lipid levels, such as nephrotic syndrome, severe liver diseases, Cushing's syndrome, or have severe arrhythmia prior to screening or randomization.
9. Poorly controlled type 2 diabetes mellitus or previously diagnosed type 1 diabetes mellitus; poorly controlled hypertension.
10. Have a history of major surgery within 3 months prior to screening, or plans to undergo major surgery during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Percentage change in mean serum triglyceride (TG) levels at Week 20 and Week 24 relative to baseline | at 20 weeks and 24 weeks of treatment

SECONDARY OUTCOMES:
Percentage change in non-HDL-C relative to baseline | at 24 weeks of treatment
Percentage change in LDL-C relative to baseline； | at 24 weeks of treatment
Percentage change in TC relative to baseline； | at 24 weeks of treatment；
Percentage change in ApoB relative to baseline； | at 24 weeks of treatment；
Percentage change in ApoA1 relative to baseline； | at 24 weeks of treatment；
Change in TG relative to baseline； | at 24 weeks of treatment；
Change in non-HDL-C relative to baseline； | at 24 weeks of treatment；
Change in LDL-C relative to baseline； | at 24 weeks of treatment；
Change in TC relative to baseline； | at 24 weeks of treatment
Change in ApoB relative to baseline； | at 24 weeks of treatment；
Change in ApoA1 relative to baseline； | at 24 weeks of treatment；
Change and percentage change in Lp(a) relative to baseline； | at 24 weeks of treatment；
Change and percentage change in HDL-C relative to baseline； | at 24 weeks of treatment；
Proportion of subjects with TG < 1.7 mmol/L； | at 24 weeks and 48 weeks of treatment；
Change and percentage change in non-HDL-C relative to baseline； | at 48 weeks of treatment；
Change and percentage change in LDL-C relative to baseline； | at 48 weeks of treatment；
Change and percentage change in TC relative to baseline； | at 48 weeks of treatment；
Change and percentage change in ApoB relative to baseline； | at 48 weeks of treatment；
Change and percentage change in ApoA1 relative to baseline； | at 48 weeks of treatment
Change and percentage change in Lp(a) relative to baseline； | at 48 weeks of treatment；
Change and percentage change in HDL-C relative to baseline； | at 48 weeks of treatment；
Change and percentage change in TG relative to baseline； | at 48 weeks of treatment；
Proportion of subjects who received rescue treatment； | Approximately a year；
Incidence and severity of adverse events and injection site reactions | Approximately a year

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided